CLINICAL TRIAL: NCT01075009
Title: Predictors of Rates of Resistant Gram-Negative Bacteria in a Consortium of Academic Medical Center Hospitals.
Brief Title: Predictors of Rates of Resistant Gram-Negative Bacteria
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: PT104983
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Relationship of Carbapenem Use to Carbapenem Resistant Gram-negative Bacteria
Keywords: Antibiotics; Resistance; Epidemiology; Gram-negative bacteria; Epidemiology of antibiotic use

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Antibiotic resistance in gram-negative bacteria continues to increase in US hospitals. This comes at a time when there are few new drugs in development that are active for these resistant organisms. The implication is that we must learn to use the drugs that we have more wisely and develop new strategies that will preserve existing agents. Antimicrobial "stewardship" programs are one strategy that many hospitals are adopting to improve the quality of antimicrobial use. The goal of this project is to develop a consortium of US academic medical centers that will allow characterization of the relationships between antibiotic use and rates of resistance for gram-negative pathogens, and to help hospital devise new strategies that will modify antibiotic use and possibly delay or reduce resistance.

The specific hypotheses are:

* Hospitals with established or emerging resistance in gram-negative pathogens, including extended spectrum beta-lactamase (ESBL) producing organisms, carbapenem-resistant enterobacteriaceae (CRE)and carbapenem-resistant P. aeruginosa have a different pattern of antimicrobial drug use compared to hospitals with fewer of these organisms.
* Hospital use of ertapenem is not associated with the rates of carbapenem-resistant organisms.

DETAILED DESCRIPTION:
Antibacterial drug use

Systemic antibacterial drug use in adult inpatients discharged between January 1, 2006 and December 31, 2010 was obtained from patient-level billing records. These data were aggregated and reported for each hospital as days of therapy per 1000 patient days (DOT/1000PD) as previously described [10]. Any dose of an antibiotic received by a patient during a 24 hour period is counted as one DOT. For example, administration of imipenem/cilastatin 1000 mg every 8 hours, or administration of 500mg every 6 hours, is counted as one DOT. We have recently reported advantages of measuring antibiotic use by DOTs versus the metric usually recommended, the Defined Daily Dose (DDD) [12].

Antimicrobial susceptibility

In year 2009 we requested the annual cumulative hospital antibiograms from the 50 hospitals for the years in which we had carbapenem drug use. The contact at each hospital was usually the antimicrobial stewardship pharmacist, but may also have included the infectious diseases physician(s), clinical microbiologist or infection control practitioner. We utilized antibiograms with a full calendar year of susceptibility reported for all clinical isolates (at least 30 isolates), the total number of isolates and the proportion of resistant isolates.

All hospitals received an on-line survey requesting additional information regarding susceptibility testing methods and antibiogram construction. We used the secure survey instruments provided by REDCap (Research electronic data capture; www.project-redcap.com) to send and compile survey responses. Specifically we inquired about the inclusion/exclusion of duplicate clinical isolates in the antibiogram, method(s) of susceptibility testing, policy regarding surveillance cultures and we attempted to verify that Clinical Laboratory Standards Institute (CLSI) interpretative breakpoints were used for all years. As recommended by Schwaber we recorded both proportions and rates of carbapenem resistant P. aeruginosa [13]. The resistant proportion was the number of resistant isolates divided by total number of isolates, and the resistant incidence rate was the number of resistant isolates per 1000 adult patient days (PD).

ELIGIBILITY:
Inclusion Criteria:

* Aggregated data from adult inpatients

Exclusion Criteria:

* Children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized adult patients
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2010-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Relationship of ertapenem use and carbapenem resistant P. aeruginosa | 2006-2011

CONTACTS AND LOCATIONS:
Overall Officials: Ron E Polk, Pharm.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Background] Pakyz AL, MacDougall C, Oinonen M, Polk RE. Trends in antibacterial use in US academic health centers: 2002 to 2006. Arch Intern Med. 2008 Nov 10;168(20):2254-60. doi: 10.1001/archinte.168.20.2254. PMID 19001203
- [Background] Pakyz AL, Oinonen M, Polk RE. Relationship of carbapenem restriction in 22 university teaching hospitals to carbapenem use and carbapenem-resistant Pseudomonas aeruginosa. Antimicrob Agents Chemother. 2009 May;53(5):1983-6. doi: 10.1128/AAC.01535-08. Epub 2009 Mar 9. PMID 19273670